CLINICAL TRIAL: NCT02355860
Title: Female Sexual Function and Socioeconomic Status
Status: Completed | Type: Observational
Sponsor: Brett Worly, MD (Other)
Responsible Party: Sponsor-Investigator, Brett Worly, MD, Primary Investigator, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 11D.84
Record Dates: First submitted 2014-11-18; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: assessment — assessment

SUMMARY:
In an urban gynecology practice serving patients with publicly and privately funded insurance, female sexual dysfunction was associated with low income, depression, urinary incontinence, and sexual inactivity.

DETAILED DESCRIPTION:
Introduction: Female sexual dysfunction is common, and the effect of socioeconomic status in an urban population is unknown. The objective is to determine socioeconomic and clinical factors associated with female sexual dysfunction for patients with publicly and privately funded health insurance in an urban outpatient gynecology clinic.

Methods: We performed an observational, IRB approved, cross-sectional study of 238 sexually-active, non-pregnant women reporting to two urban gynecology clinics, representing patients with publicly funded (n=70) or privately funded health insurance (n=168). The participants completed validated questionnaires measuring sexual function (Female Sexual Function Index or FSFI), depression (Center for Epidemiologic Studies Depression Scale), urinary incontinence (Questionnaire for Urinary Incontinence Diagnosis), and demographic variables. Data was analyzed with non-parametric t-tests, chi-squared tests, and linear regression models.

ELIGIBILITY:
Inclusion Criteria:

* women age 18 or older, presenting for an annual routine gynecology appointment, and were sexually active in the past six months

Exclusion Criteria:

* pregnant women, women who were less than six weeks post-partum, women reporting for a gynecologic problem visit, non-English speakers, incomplete survey questionnaires, or refusal to consent to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 238 sexually-active, non-pregnant women reporting to two urban gynecology clinics, representing patients with publicly funded (n=70) or privately funded health insurance (n=168).
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
FSF Index | Day 1
  Questionnaire

SECONDARY OUTCOMES:
Health Information Assessment | Day 1
  Questionnaire